CLINICAL TRIAL: NCT06918210
Title: Indocyanine Green Fluorescence During Fundus First Laparoscopic Cholecystectomy
Acronym: INFUNDUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Västernorrland (Unknown)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INFUNDUS
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Gallstone; Gallstone; Cholecystitis, Acute
Keywords: cholecystectomy; Indocyanine Green; Bile duct injury; Intraoperative cholangiography; Fundus first
MeSH Terms: conditions — Gallstones; Cholecystitis | interventions — Indocyanine Green

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visualization with ICG (Experimental): Intraoperative visualization of the bile ducts with ICG and near infrared light
  Interventions: Procedure: Indocyanine Green; Procedure: Cholangiography
- Comparator (Active Comparator): Visualization of the bile ducts with intraoperative cholangiography only.
  Interventions: Procedure: Cholangiography

INTERVENTIONS:
Procedure: Indocyanine Green — Visualization of the bile ducts with ICG
  Arms: Visualization with ICG
Procedure: Cholangiography — Visualization of the bile ducts with intraoperative cholangiography

SUMMARY:
Laparoscopic cholecystectomy is the routine method for managing gallstone disease. This is considered a safe procedure with low risk of severe complications. Lesions to the deep bile ducts is, however, a rare complication from laparoscopic cholecystectomy that may have devastating consequences. The risk of bile duct injuries may be reduced by adapting the surgical approach. In general, the operation is started from the lower part of the gallbladder and continued upwards. It may, however, also be initiated from the top of the gallbladder and extended downwards. This approach, also termed fundus first, is routine at a few units.

By injecting Indocyanin Green (ICG) that is excreted into the bile, the bile ducts may be visualized using near infrared light. This is a technique for mapping the anatomical structures adjacent to the gallbladder that has been used in previous studies for preventing bile duct injuries. This method has, however, not been tested at units where fundus first is the routine surgical technique. In the present randomized controlled trial, the investigators intend to evaluate the safety of ICG as a means for reducing the risk of bile duct lesions and to see if it works as intended.

Altogether 294 operations for gallstones will be included in the study. The patients will be randomized to surgery with or without ICG. Regardless of the randomization, all operations will be undertaken with the fundus first technique.

Thirty days after the operation, all data related to the operation are retrieved from the patient records by an assessor that does not know what group the patient was randomized to. The primary endpoint of the study is the time required from the start of the operation until intraoperative cholangiography is done. In addition, total operative time, all surgical complications and need for converting the operation to an open procedure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* Verbal and written consent provided
* Age ≥ 18 years

Exclusion Criteria:

* Thyroid disease
* Allergy against ICG or Iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to intraoperative cholangiography | During procedure.
  Time from first incision until intraoperative cholangiography

SECONDARY OUTCOMES:
Procedure-related complications | Up to 30 days postoperatively
  Complications related to the cholecystectomy confirmed intraoperatively or postoperatively
Total operative time | During procedure
  Time from first incision to closure of the wounds
Intraoperative gallbladder perforation | During procedure
  Intraoperative iatrogenic gallbladder perforation
Conversion from laparoscopic to open cholecystectomy | During procedure
  Decision to convert from laparoscopic to open cholecystectomy taken intraoperatively
Surgeon perception of complexity | During procedure
  The perception of the complexity of the procedure rated by the surgeon on a numeric rating scale from 0 to 10 where 10 indicates the highest level of complexity
Patient reported outcome | Up to 30 days postoperatively
  Symptoms and satisfaction rated by the patient 30 days postoperatively on a numeric rating scale from 0 to 10 where 10 indicates the highest level of satisfaction and absence of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yucel Cengiz, MD, PhD, Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: Yes
Data related to the study may be shared on request to the principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2026 to December 2030
URL: https://ki.se/ki-sos/gastrointestinal-kirurgi-ki-sos/regionalt-natverk-for-studier-av-benign-hpb-kirurgi